CLINICAL TRIAL: NCT05410132
Title: Internet-based Mindfulness-based Training (iMBT) for People With Depression: Investigation of Its Efficacy and Mechanism of Change
Brief Title: Internet-based Mindfulness-based Training (iMBT) for People With Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Winnie W.S. MAK, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SBRE-21-0158
Record Dates: First submitted 2022-05-26; First posted 2022-06-08 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Mindfulness; Depression
Keywords: mental well-being; depression; Internet-based Mindfulness-based Training; online
MeSH Terms: conditions — Depression; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internet-based mindfulness-based training group (iMBT) (Experimental): Participants in the iMBT group will be expected to complete an Internet-based mindfulness-based training delivered over a 6-week period via an internet e-learning mental health platform. They will be assessed at four different time points:
  (1) before intervention (T0), (2) 2,4 weeks since the commencement of group (T1,2), (3) 6 weeks after (i.e., when the intervention ends) (T3), (4) at 3-month follow-up(T4).
  Interventions: Other: Internet-delivered Mindfulness Based Training (iMBT)
- Treatment-as-usual control group (TAU) (No Intervention): The TAU group will be advised to seek assistance from their usual healthcare provider when needed. They will be offered access to the Internet-based mindfulness-based course content after the study has ended.

INTERVENTIONS:
Other: Internet-delivered Mindfulness Based Training (iMBT) — The iMBT developed for this study will be adapted from our team's previous study and the manual of mindfulness based cognitive therapy. The program is designed to be brief in nature, for example, participants will be asked to practice meditations for 15 minutes a day instead of the original 45 minutes a day, and each module is shortened to approximately 1 hour instead of the original 2.5 hours.
  This iMBT is comprised of six weekly modules on education about mindfulness, guidance on using mindfulness skills to manage symptoms, guided meditations (e.g., mindful breathing, mindful eating, mindful walking, body scan, acceptance, choiceless awareness and disengaging from thoughts exercise), and guidance on using informal mindfulness skills in day-to-day life. Readings, audio and graphics are included to explain the concept of mindfulness and overcome common difficulties associated with mindfulness practice.
  Arms: Internet-based mindfulness-based training group (iMBT)

SUMMARY:
The research goals of this randomized controlled trial are to determine the feasibility and the mechanism of change of iMBT that has been developed using the Acceptance Checklist for Clinical Effectiveness Pilot Trials.

The primary research question is as follows:

What is the effectiveness of the iMBT in relation to improvements on depressive symptoms among people with clinical depression, relative to a usual care control after the intervention and in 3-month follow-up?

Secondary questions include the following:

Which facet(s) of mindfulness (i.e., observe, describe, act with awareness, non-react and non-judgement) improved during the intervention? How does the growth trajectory of different facets of mindfulness relate to the improvement of well-being and reduction of ill-being?

The investigators hypothesize that:

H1 Participants in iMBT group will have greater reduction in depressive symptoms and increase in all facets of mindfulness and mental well-being, than the usual care group at post-intervention, and 3-month follow-up.

H2 Using latent growth analysis, the intraindividual growth trajectory of the monitor and acceptance facets of mindfulness would mediate the effect of iMBT on the intraindividual changes in depressive symptoms.

H3 Using multi-group analysis, in accord with Acceptance and Monitor theory, the relationship between the growth trajectory of monitor facets of mindfulness and the growth trajectory of depressive symptoms will be moderated by the level of acceptance. People with greater acceptance of inner experience will benefit more from the change of monitor facets of mindfulness in iMBT.

DETAILED DESCRIPTION:
1.1 Internet delivered Intervention for Depression Major depressive disorder (MDD) is a significant and common public health concern due to its high prevalence, high disease burden, and common comorbidity 1-3. While evidence-based psychological treatments are available, most of those affected by depression do not have access to these treatments or seek help5. Several reasons such as long waiting time of mental health service, barriers in access to care, and reluctance to seek help due to stigma are contributing to this situation6. One promising approach to enhance the accessibility and serviceability of psychotherapy is to complement the existing system using evidence-based self-management programs delivered via the Internet. Different forms of psychotherapy, could potentially be transferable to Internet-based interventions, especially when guided by coaches9 who provide online guidance, encouragement, and therapeutic activities 10,11. The initiatives of translating and scaling up mental health service via the Internet echo with the National Institute for Health and Care Excellence guidelines (NICE) for managing depression 12. The guideline recommended low-intensity Internet-based interventions as first line treatment prior to more complex higher-tier services. Internet-based interventions for major depression has not only been shown to be efficacious 13, but also cost-effective and able to generate societal savings14,15. Notably, a recent meta-analytic review revealed that Internet-based cognitive behavioral therapy (iCBT) was as effective as its face-to-face counterpart for clinical practice in treating depression16. Given the high accessibility and low recurring costs of Internet-based interventions for depression, these interventions are suggested to have a huge potential for public mental health impact.

1.2 Mindfulness-based Training as an Internet delivered Intervention for People with Depression In addition to iCBT, Internet-based mindfulness-based training (iMBT) has also gained evidence in improving mental well-being and reducing psychological distress. Mindfulness is defined "paying attention in a particular way: on purpose, in the present moment, and nonjudgmentally" 17,18. In the context of understanding the beneficial effect of mindfulness on depression, it is theorized that mindfulness training reduced depression through encouraging individuals to notice experiences regardless of its valence labelled, and to approach those experiences with gentleness, curiosity and interest without suppressing, judging, or pushing these experiences away 19. In turn, repetitive negative thinking, which involves cognitive over-engagement in attempt to control unpleasant inner experiences, would be attenuated by the facilitation of individuals' processing of their affective experiences17,20. Moreover, through observing that different experiences come and go over time, mindfulness practitioners come to know the impermanent and transitory nature of the inner experience and realize that it is not always necessary to react.

A recent meta-analysis that included 209 studies with 12,145 participants concluded that mindfulness-based intervention is an effective treatment for various psychological problems, and is especially effective for reducing depression, anxiety and stress21. Evidence of online mindfulness-based intervention has demonstrated its effectiveness among community samples and subclinical populations with elevated depressive symtoms23,24. In addition, iMBT may be more acceptable than intervention using the traditional cognitive behavioral approach. As reported in a recent study, intervention with mindfulness element was chosen as the first option of intervention by over 80% of people with depression/anxiety. Moreover, nearly half of the participants in a study reported preference of online formats for mindfulness interventions over group/individual formats28.

Given its acceptability and preference by individuals with mental health needs and its promising effects in reducing depressive and anxiety symptoms, another critical question lies in examining how MBT works so that further refinement of such approach can be made based on its theoretical roots and mechanism of change. The precise mechanisms underlying the effect of mindfulness have received recent theoretical attention19,29,30. Despite not having abundant studies, recent meta-analysis of mediation studies with 12 RCTs identified consistent evidence for the change in mindfulness as a mechanism underlying MBIs31. However, simply identifying mindfulness as the mechanism of change in MBT is too crude and intuitive. Further unpacking the effects of mindfulness is necessary to understand the process through which individuals experience changes. One possibility is to examine specific effect of each facet in mindfulness (i.e., observe, describe, act with awareness, non-react and non-judgement). Correlational study suggested that different facets of mindfulness have differential relationships with various psychological variables 32. Although most facets of mindfulness are frequently found to be associated with reduced psychological distress, the "observe" facets is often uncorrelated or even positively correlated with mood symptoms 33. In accord with the Acceptance and Monitor theory19, a recent study showed high observing skills was correlated with higher depressive symptoms with low acceptance. Yet, high observing skills in combination with high acceptance correlated with increased adaptive cognitive processing tendencies 34. Consequently, it is important to examine relationships between change of mindfulness and that of psychological symptoms at the facet level to provide a more fine-grained perspective on the contribution of mindfulness. This could also facilitate refinement of iMBT.

1.3 Aims and hypotheses The research goals of this randomized controlled trial are to determine the feasibility and the mechanism of change of iMBT that has been developed using the Acceptance Checklist for Clinical Effectiveness Pilot Trials (ACCEPT) framework35.

The primary research question is as follows:

What is the effectiveness of the iMBT in relation to improvements on depressive symptoms among people with clinical depression, relative to a usual care control after the intervention and in 3-month follow-up?

Secondary questions include the following:

Which facet(s) of mindfulness (i.e., observe, describe, act with awareness, non-react and non-judgement) improved during the intervention? How does the growth trajectory of different facets of mindfulness relate to the improvement of well-being and reduction of ill-being?

The investigators hypothesize that:

H1 Participants in iMBT group will have greater reduction in depressive symptoms and increase in all facets of mindfulness and mental well-being, than the usual care group at post-intervention, and 3-month follow-up.

H2 Using latent growth analysis, the intraindividual growth trajectory of the monitor and acceptance facets of mindfulness would mediate the effect of iMBT on the intraindividual changes in depressive symptoms.

H3 Using multi-group analysis, in accord with Acceptance and Monitor theory, the relationship between the growth trajectory of monitor facets of mindfulness and the growth trajectory of depressive symptoms will be moderated by the level of acceptance. People with greater acceptance of inner experience will benefit more from the change of monitor facets of mindfulness in iMBT.

A two-armed parallel RCT following CONSORT statement1 will be conducted to examine the efficacy of an Internet-based mindfulness-based training (iMBT) to a treatment-as-usual control group (TAU). Eligible participants will be randomized to either iMBT or TAU by block randomization with block number of 6 with allocation ratio of 1:1. Intervention (iMBT) will be delivered over a 6-week period via an internet e-learning mental health platform. Both groups will be assessed at the following time points: (1) before intervention (T0), (2) 2,4 weeks since the commencement of group (T1,2), (3) 6 weeks after (i.e., when the intervention ends) (T3), (4) at 3-month follow-up(T4).

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 18 years old or above
* Have access to computer and mobile phone (since this is an internet-based therapy)
* Score >9 on PHQ9
* Have the ability to read and type Chinese

Exclusion Criteria:

* Self-reported presence of psychosis or bipolar disorder, post-traumatic stress disorder, drug or alcohol dependence, current use of antipsychotic medications
* Self-reported frequent suicidal ideation (more than half of the days in the past two weeks)
* Completion of an online mental health program/research for depression in the past 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2022-03-24 (Actual); Primary Completion 2024-03-30 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
Depression | at baseline
  Patient Health Questionnaire (PHQ9) (Kroenke, Spitzer, & Williams, 2001). It is a 9-item measure to access the severity of depression. PHQ-9 has been validated and used widely in the general population for screening and measuring depression severity. Scores of 5, 10, 15, and 20 denote mild, moderate, moderately severe, and severe level of depression respectively (range: 0-27).
Depression | 2nd week
  Patient Health Questionnaire (PHQ9) (Kroenke, Spitzer, & Williams, 2001). It is a 9-item measure to access the severity of depression. PHQ-9 has been validated and used widely in the general population for screening and measuring depression severity. Scores of 5, 10, 15, and 20 denote mild, moderate, moderately severe, and severe level of depression respectively (range: 0-27).
Depression | 4th week
  Patient Health Questionnaire (PHQ9) (Kroenke, Spitzer, & Williams, 2001). It is a 9-item measure to access the severity of depression. PHQ-9 has been validated and used widely in the general population for screening and measuring depression severity. Scores of 5, 10, 15, and 20 denote mild, moderate, moderately severe, and severe level of depression respectively (range: 0-27).
Depression | 6th week
  Patient Health Questionnaire (PHQ9) (Kroenke, Spitzer, & Williams, 2001). It is a 9-item measure to access the severity of depression. PHQ-9 has been validated and used widely in the general population for screening and measuring depression severity. Scores of 5, 10, 15, and 20 denote mild, moderate, moderately severe, and severe level of depression respectively (range: 0-27).
Depression | 18th week
  Patient Health Questionnaire (PHQ9) (Kroenke, Spitzer, & Williams, 2001). It is a 9-item measure to access the severity of depression. PHQ-9 has been validated and used widely in the general population for screening and measuring depression severity. Scores of 5, 10, 15, and 20 denote mild, moderate, moderately severe, and severe level of depression respectively (range: 0-27).

SECONDARY OUTCOMES:
Mindfulness | at baseline, 2nd, 4th, 6th, and 18th week
  Five Facets Mindfulness Questionnaire - Short form (FFMQ-SF) (Hou et al., 2013). It is a 20-item measure that examines the five facets of mindfulness, namely, observe, describe, act with awareness, non-judging of inner experience, and non-reactivity to inner experience.
Mental Well-being | at baseline, 2nd, 4th, 6th, and 18th week
  The Warwick Edinburgh Mental Well-being Scale (Tennant et al, 2007) WEMWBS is a measure of mental well-being focusing entirely on positive aspects of mental health. It is a 7-item measure, using a 5-point Likert scale from 1 (none of the time) to 5 (all of the time).
Credibility and Expectancy | at baseline, 2nd, 4th, 6th, and 18th week
  The Credibility and Expectancy Questionnaire (CEQ) (Devilly & Borkovec, 2000) is a 6-item measure, using a scale from 0% to 100%.
Difficulties in Emotional Regulation Scale | at baseline, 2nd, 4th, 6th, and 18th week
  The Difficulties in Emotional Regulation Scale (DERS) is a 16-item measure focusing on emotion regulation. Items are rated on a scale of ("almost never [0-10%]") to ("almost always [91-100%]"). Higher scores indicate more difficulty in emotion regulation.
Non-attachment | at baseline, 2nd, 4th, 6th, and 18th week
  The Nonattachment Scale-Short Form (Chio, Lai, & Mak, 2018) was used to measure nonattachment. Participants rated the items from 1 (disagree strongly) to 6 (agree strongly). Excellent internal consistency was demonstrated in the previous studies.
Stillness | at baseline, 2nd, 4th, 6th, and 18th week
  Stillness scale is a 13-item measure focusing on stillness.
Equanimity | at baseline, 2nd, 4th, 6th, and 18th week
  The Equanimity Barriers Scale (Juneau, Pellerin, Trives, Ricard, Shankland & Dambrun, 2020) was used. This instrument is a 14-item self-report questionnaire to measure barriers that individuals encounter in developing equanimity, rather than an individual's degree of equanimity.
Peace of mind | at baseline, 2nd, 4th, 6th, and 18th week
  Peace of mind was measured using the Peace of mind scale. Participants were asked to indicate their internal state of peacefulness and harmony, using a scale of 1 (never) to 5 (always).

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychology, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ferrari AJ, Somerville AJ, Baxter AJ, Norman R, Patten SB, Vos T, Whiteford HA. Global variation in the prevalence and incidence of major depressive disorder: a systematic review of the epidemiological literature. Psychol Med. 2013 Mar;43(3):471-81. doi: 10.1017/S0033291712001511. Epub 2012 Jul 25. PMID 22831756
- [Background] Liu Q, He H, Yang J, Feng X, Zhao F, Lyu J. Changes in the global burden of depression from 1990 to 2017: Findings from the Global Burden of Disease study. J Psychiatr Res. 2020 Jul;126:134-140. doi: 10.1016/j.jpsychires.2019.08.002. Epub 2019 Aug 10. PMID 31439359
- [Background] Patel V, Chisholm D, Parikh R, Charlson FJ, Degenhardt L, Dua T, Ferrari AJ, Hyman S, Laxminarayan R, Levin C, Lund C, Medina Mora ME, Petersen I, Scott J, Shidhaye R, Vijayakumar L, Thornicroft G, Whiteford H; DCP MNS Author Group. Addressing the burden of mental, neurological, and substance use disorders: key messages from Disease Control Priorities, 3rd edition. Lancet. 2016 Apr 16;387(10028):1672-85. doi: 10.1016/S0140-6736(15)00390-6. Epub 2015 Oct 8. PMID 26454360
- [Background] Russ TC, Stamatakis E, Hamer M, Starr JM, Kivimaki M, Batty GD. Association between psychological distress and mortality: individual participant pooled analysis of 10 prospective cohort studies. BMJ. 2012 Jul 31;345:e4933. doi: 10.1136/bmj.e4933. PMID 22849956
- [Background] Kazdin AE. Addressing the treatment gap: A key challenge for extending evidence-based psychosocial interventions. Behav Res Ther. 2017 Jan;88:7-18. doi: 10.1016/j.brat.2016.06.004. PMID 28110678
- [Background] Magaard JL, Seeralan T, Schulz H, Brutt AL. Factors associated with help-seeking behaviour among individuals with major depression: A systematic review. PLoS One. 2017 May 11;12(5):e0176730. doi: 10.1371/journal.pone.0176730. eCollection 2017. PMID 28493904
- [Background] Andersson G, Titov N. Advantages and limitations of Internet-based interventions for common mental disorders. World Psychiatry. 2014 Feb;13(1):4-11. doi: 10.1002/wps.20083. PMID 24497236
- [Background] Fairburn CG, Patel V. The impact of digital technology on psychological treatments and their dissemination. Behav Res Ther. 2017 Jan;88:19-25. doi: 10.1016/j.brat.2016.08.012. PMID 28110672
- [Background] Johansson R, Andersson G. Internet-based psychological treatments for depression. Expert Rev Neurother. 2012 Jul;12(7):861-9; quiz 870. doi: 10.1586/ern.12.63. PMID 22853793
- [Background] Andersson G, Carlbring P, Titov N, Lindefors N. Internet Interventions for Adults with Anxiety and Mood Disorders: A Narrative Umbrella Review of Recent Meta-Analyses. Can J Psychiatry. 2019 Jul;64(7):465-470. doi: 10.1177/0706743719839381. Epub 2019 May 16. PMID 31096757
- [Background] Donker T, Blankers M, Hedman E, Ljotsson B, Petrie K, Christensen H. Economic evaluations of Internet interventions for mental health: a systematic review. Psychol Med. 2015 Dec;45(16):3357-76. doi: 10.1017/S0033291715001427. Epub 2015 Aug 3. PMID 26235445
- [Background] Tate DF, Finkelstein EA, Khavjou O, Gustafson A. Cost effectiveness of internet interventions: review and recommendations. Ann Behav Med. 2009 Aug;38(1):40-5. doi: 10.1007/s12160-009-9131-6. PMID 19834778
- [Background] Andersson G, Topooco N, Havik O, Nordgreen T. Internet-supported versus face-to-face cognitive behavior therapy for depression. Expert Rev Neurother. 2016;16(1):55-60. doi: 10.1586/14737175.2015.1125783. Epub 2015 Dec 15. PMID 26610160
- [Background] Chambers R, Gullone E, Allen NB. Mindful emotion regulation: An integrative review. Clin Psychol Rev. 2009 Aug;29(6):560-72. doi: 10.1016/j.cpr.2009.06.005. Epub 2009 Jun 23. PMID 19632752
- [Background] Lindsay EK, Creswell JD. Mechanisms of mindfulness training: Monitor and Acceptance Theory (MAT). Clin Psychol Rev. 2017 Feb;51:48-59. doi: 10.1016/j.cpr.2016.10.011. Epub 2016 Nov 5. PMID 27835764
- [Background] Lang AJ. What mindfulness brings to psychotherapy for anxiety and depression. Depress Anxiety. 2013 May;30(5):409-12. doi: 10.1002/da.22081. Epub 2013 Feb 19. No abstract available. PMID 23423991
- [Background] Khoury B, Lecomte T, Fortin G, Masse M, Therien P, Bouchard V, Chapleau MA, Paquin K, Hofmann SG. Mindfulness-based therapy: a comprehensive meta-analysis. Clin Psychol Rev. 2013 Aug;33(6):763-71. doi: 10.1016/j.cpr.2013.05.005. Epub 2013 Jun 7. PMID 23796855
- [Background] Boggs JM, Beck A, Felder JN, Dimidjian S, Metcalf CA, Segal ZV. Web-based intervention in mindfulness meditation for reducing residual depressive symptoms and relapse prophylaxis: a qualitative study. J Med Internet Res. 2014 Mar 24;16(3):e87. doi: 10.2196/jmir.3129. PMID 24662625
- [Background] Spijkerman MP, Pots WT, Bohlmeijer ET. Effectiveness of online mindfulness-based interventions in improving mental health: A review and meta-analysis of randomised controlled trials. Clin Psychol Rev. 2016 Apr;45:102-14. doi: 10.1016/j.cpr.2016.03.009. Epub 2016 Apr 1. PMID 27111302
- [Background] Pots WT, Meulenbeek PA, Veehof MM, Klungers J, Bohlmeijer ET. The efficacy of mindfulness-based cognitive therapy as a public mental health intervention for adults with mild to moderate depressive symptomatology: a randomized controlled trial. PLoS One. 2014 Oct 15;9(10):e109789. doi: 10.1371/journal.pone.0109789. eCollection 2014. PMID 25333885
- [Background] Hofmann SG, Sawyer AT, Witt AA, Oh D. The effect of mindfulness-based therapy on anxiety and depression: A meta-analytic review. J Consult Clin Psychol. 2010 Apr;78(2):169-83. doi: 10.1037/a0018555. PMID 20350028
- [Background] Barth J, Munder T, Gerger H, Nuesch E, Trelle S, Znoj H, Juni P, Cuijpers P. Comparative efficacy of seven psychotherapeutic interventions for patients with depression: a network meta-analysis. PLoS Med. 2013;10(5):e1001454. doi: 10.1371/journal.pmed.1001454. Epub 2013 May 28. PMID 23723742
- [Background] Wahbeh H, Svalina MN, Oken BS. Group, One-on-One, or Internet? Preferences for Mindfulness Meditation Delivery Format and their Predictors. Open Med J. 2014;1:66-74. doi: 10.2174/1874220301401010066. Epub 2014 Nov 28. PMID 27057260
- [Background] Teper R, Inzlicht M. Meditation, mindfulness and executive control: the importance of emotional acceptance and brain-based performance monitoring. Soc Cogn Affect Neurosci. 2013 Jan;8(1):85-92. doi: 10.1093/scan/nss045. Epub 2012 Apr 15. PMID 22507824
- [Background] Gu J, Strauss C, Bond R, Cavanagh K. How do mindfulness-based cognitive therapy and mindfulness-based stress reduction improve mental health and wellbeing? A systematic review and meta-analysis of mediation studies. Clin Psychol Rev. 2015 Apr;37:1-12. doi: 10.1016/j.cpr.2015.01.006. Epub 2015 Jan 31. PMID 25689576

DOCUMENTS (1):
  • Study Protocol (2021-09-24): https://cdn.clinicaltrials.gov/large-docs/32/NCT05410132/Prot_001.pdf